CLINICAL TRIAL: NCT07001462
Title: Effects of Combined Inspiratory Muscle Training and Positive Expiratory Pressure Therapy on Pulmonary Function, Respiratory Muscle Strength, Exercise Capacity and Dyspnea in Stable Group E COPD Patients
Brief Title: Effectiveness of IMT/PEP Therapy in Group E COPD and Comparison of GOLD vs STAR Classifications
Status: Completed | Type: Observational
Sponsor: Bugra Kerget (Other)
Responsible Party: Sponsor-Investigator, Bugra Kerget, Asc.Prof.Dr., Ataturk University
Organization: Ataturk University (Other)
Other Study IDs: B.30.2ATA.0.01.00/487; BAP-13001 (Atatürk University) (Other Grant/Funding Number: Atatürk University)
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: COPD; Inspiratory Muscle Training
Keywords: COPD; inspiratory muscle training; pulmonary rehabilitation; GOLD; STAR
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IMT/PEP Group: Patients with Group E chronic obstructive pulmonary disease (COPD) who received standardized pharmacological treatment combined with inspiratory muscle training and positive expiratory pressure (IMT/PEP) therapy. The intervention was administered using a dual-function device twice daily for 12 weeks.
  Interventions: Behavioral: Inspiratory Muscle Training / Positive Expiratory Pressure (IMT/PEP) Therapy

INTERVENTIONS:
Behavioral: Inspiratory Muscle Training / Positive Expiratory Pressure (IMT/PEP) Therapy — IMT/PEP therapy was administered using a dual-function device (BİO Breathe, Korea) designed to provide both inspiratory muscle resistance and positive expiratory pressure. Patients performed the therapy for 15 minutes, twice daily, over a 12-week period, in addition to standard pharmacological treatment. Pressure levels were individually adjusted between 5-40 cmH₂O based on patient capacity.

SUMMARY:
Background:

Inspiratory muscle training combined with positive expiratory pressure (IMT/PEP) may improve outcomes in chronic obstructive pulmonary disease (COPD), but evidence in exacerbation-prone (Group E) disease is limited. This study is designed to evaluate the effects of IMT/PEP on pulmonary function, respiratory muscle strength, exercise capacity, and dyspnea in stable Group E COPD.

Methods :

This prospective randomized controlled trial will enroll 62 patients with stable Group E COPD between June 2023 and September 2024. Participants will be randomized to receive IMT/PEP plus standard care or standard care alone. Pulmonary function tests, maximal inspiratory pressure (MIP), maximal expiratory pressure (MEP), six-minute walk test (6MWT), oxygen saturation (SO₂), and dyspnea scales (mMRC, CAT, MBS, VAS) will be assessed at baseline, 1 month, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 40 years

Diagnosis of Group E COPD according to GOLD 2023 criteria

Post-bronchodilator FEV₁/FVC < 0.70 and FEV₁ < 50% predicted

mMRC score ≥ 2 or CAT score ≥ 10

History of ≥2 exacerbations or ≥1 hospitalization in the past year

Stable clinical condition (no exacerbation in the past 2 weeks)

Ability and willingness to perform IMT/PEP therapy

Provided written informed consent

Exclusion Criteria:

Acute exacerbation of COPD at time of enrollment

Contraindications to pulmonary function testing or 6-minute walk test (e.g., recent myocardial infarction, unstable angina)

Inability to perform inspiratory or expiratory maneuvers reliably (e.g., due to cognitive or neuromuscular disorders)

Significant orofacial muscle weakness unresponsive to modified mouthpiece

Participation in another interventional study within the past 3 months

Nonadherence to COPD treatment plan

Any condition deemed by investigators to interfere with study participation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 40 years and older diagnosed with Group E chronic obstructive pulmonary disease (COPD) according to GOLD 2024 criteria, with moderate to very severe airflow limitation, increased symptom burden, and a history of frequent exacerbations or hospitalizations.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Change in Maximal Inspiratory Pressure (MIP) After 12 Weeks of IMT/PEP Therapy | Baseline and Week 12
  Maximal inspiratory pressure (MIP) was measured at baseline and after 12 weeks using a digital manometer at residual volume (RV) to evaluate the effect of IMT/PEP therapy on inspiratory muscle strength.
Change in Residual Volume (RV) After 12 Weeks of IMT/PEP Therapy | Baseline and Week 12
  Residual volume (RV) was obtained through whole-body plethysmography at baseline and after 12 weeks to assess the impact of IMT/PEP therapy on pulmonary hyperinflation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. Data sharing may be considered upon reasonable request, pending ethical approval and institutional data protection policies.